CLINICAL TRIAL: NCT01477723
Title: Evaluation of an Oral Nutritional Supplement Containing AN 777 in Older Hospitalized Patients
Brief Title: Evaluation of an Oral Nutritional Supplement in Older Hospitalized Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BK33
Record Dates: First submitted 2011-11-19; First posted 2011-11-22 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental Oral Nutrition Supplement (Experimental): Experimental ONS orally Two 8 fl oz servings/day
  Interventions: Other: Experimental Oral Nutritional Supplement
- No Product (No Intervention)

INTERVENTIONS:
Other: Experimental Oral Nutritional Supplement — Experimental ONS orally Two 8 fl oz servings/day
  Arms: Experimental Oral Nutrition Supplement

SUMMARY:
Study objectives are to verify the loss of lean mass during a hospital stay in a group of older patients; to evaluate the effects of consuming a high-calorie complete and balanced oral nutritional supplement; to collect post-discharge information.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 55 years of age.
2. Admitted to hospital with a disease of respiratory system including acute respiratory diseases (e.g., pneumonia, acute bronchitis) or exacerbation of existing respiratory diseases.
3. Anticipated length of hospital stay of at least 3 days.
4. Ability to climb a flight of 10 stairs or walk a city block without the help of another person prior to hospitalization.
5. Able to consume foods and beverages orally.

Exclusion Criteria:

1. Unstable heart failure which requires ICU admission.
2. Severe respiratory disease requiring long-term, continuous oxygen therapy.
3. Diabetes.
4. Impaired renal function.
5. Impaired liver function.
6. Cancer.
7. Hospitalized for two or more days in past 4 weeks.
8. Requires intubation or tube feeding.
9. Expected to be transferred to an advanced care unit.
10. Body mass index of ≥ 40 kg/m2.
11. Active tuberculosis.
12. Ascites or severe edema.
13. Acute Hepatitis or HIV.
14. Disorder of gastrointestinal tract.
15. Dementia;brain metastases, eating disorder, significant neurological, psychiatric disorder, other psychological condition.
16. Medication/dietary supplements/substances that could modulate metabolism or weight.
17. Partial or full artificial lower limb.
18. Allergy or intolerance to any of the ingredients in the study products.
19. Procedure using iodine-based contrast media within 7 days prior to hospitalization; or, anticipated to need procedure using iodine-based contrast media within 3 days after hospital admission.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Leg Lean Mass | baseline to day 30

SECONDARY OUTCOMES:
Body Weight | baseline to day 30
Body Mass Index | baseline to day 30
Activities of daily living | baseline to day 30

CONTACTS AND LOCATIONS:
Overall Officials: Vikkie Mustad, PhD, Study Chair — Abbott Nutrition
Locations (14):
- United States (12):
  - Horizon Research Group Inc, Mobile, Alabama
  - Northwestern University, Chicago, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Central Maine Medical Center, Lewiston, Maine
  - William Beaumont Hospital, Royal Oak, Michigan
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Mount Carmel West Hospital, Columbus, Ohio
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas Medical Branch, Galveston, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Salem VA Medical Center, Salem, Virginia
- Puerto Rico (2):
  - Hospital HIMA San Pablo, Bayamón, Puerto Rico
  - Manati Medical Center, Manatí, Puerto Rico